CLINICAL TRIAL: NCT04305925
Title: Office-based Focal Laser Ablation of Prostate Cancer: An Early Feasibility Study Using MRI/US Image Fusion for Guidance
Brief Title: Focal Laser Ablation of Prostate Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-001502; 5R01CA218547 (NIH)
Record Dates: First submitted 2020-03-06; First posted 2020-03-12 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: prostrate; ablation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an open-label early feasibility/pilot study to evaluate the safety and feasibility of the focal laser ablation (FLA) Orion System. Men with histologically confirmed, non-metastatic, prostate adenocarcinoma, clinical stage ≤ T2b, with Gleason score 7 by MRI-ultrasound fusion targeted biopsy, without history of prior treatment and without neoadjuvant radiation or hormone therapy, who desire focal treatment with laser ablation will be enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Focal Laser Ablation (Experimental): The Orion system will be used to deploy and monitor thermal energy in cancerous regions of the prostate, identified by MRI and confirmed by targeted biopsy.
  Interventions: Device: Focal Laser Ablation

INTERVENTIONS:
Device: Focal Laser Ablation — Orion system to deploy and monitor thermal energy in cancerous regions of the prostate, identified by MRI and confirmed by targeted biopsy. MRI guidance will be achieved by MRI/ultrasound fusion, overlaying stored MRI images upon real-time ultrasound images. Interstitial laser treatments would be achieved by inserting the fiber into the cancerous regions guided by the Artemis image-fusion device. Applications of laser energy up to 15 watts of power will be used to treat the target region.

SUMMARY:
The primary objective of this study is to evaluate the safety and feasibility of Magnetic-Resonance(MR)-ultrasound image fusion-guided transrectal-based focal laser ablation (FLA) of prostate cancer using the Orion System, an investigational laser-based interstitial irradiation/thermal soft-tissue ablation system. Safety and feasibility will be determined by analyzing the number, type, and severity of adverse events.

DETAILED DESCRIPTION:
The primary objective is to evaluate the safety and feasibility of MR-ultrasound image fusion-guided transrectal-based focal laser ablation (FLA) of prostate cancer using the Orion System, an investigational laser-based interstitial irradiation/thermal soft-tissue ablation system. Safety and feasibility will be determined by analyzing the number, type, and severity of adverse events. In addition, changes in health-related quality of life (HRQOL) will be evaluated using Expanded Prostate Index Composite for Clinical Practice (EPIC-CP), Memorial Anxiety Scale for Prostate Cancer (MAX-PC), and Decision Regret Scale.

This is an open-label early feasibility/pilot study to evaluate the safety and feasibility of the Orion System. In this study, the investigators intend to use the investigational Orion system to deploy and monitor thermal energy in cancerous regions of the prostate, identified by MRI and confirmed by targeted biopsy. MRI guidance will be achieved by MRI/ultrasound fusion, overlaying stored MRI images upon real-time ultrasound images. Interstitial laser treatments would be achieved by inserting the fiber into the cancerous regions guided by the Artemis image-fusion device. Applications of laser energy up to 15 watts of power will be used to treat the target region. Subjects will return to clinic 1 week, 1 month, and every 3 months until one year post-FLA to be monitored for adverse events and complete Health Related Quality of Life (HRQOL) questionnaires. Biomarker (PSA) kinetics will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with untreated, organ-confined prostate cancer (clinical stage ≤ T2b, Gleason =7) x Age 40 to 85 years of age
* Multi-parametric MRI at University of California at Los Angeles (UCLA) within 6 months of study treatment, demonstrating a Region of interest (ROI) of MRI (PIRADSv2 > Grade 3). x Prostate volume 20cc to 80cc
* Transrectal ultrasound-guided biopsy with ≥ 10 systematic biopsy cores and ≥ 2 targeted biopsy cores from above MRI-derived ROI within 6 month of biopsy results
* Histologically-confirmed adenocarcinoma from targeted biopsy cores x Overall Gleason = 3+4 or 4+3
* Subjects desire focal therapy and decline conventional treatment (active surveillance, radical prostatectomy, radiation therapy, cryosurgery and hormone therapy)
* Signed informed consent for the FLA treatment through the 12 month follow-up

Exclusion Criteria:

* Any significant cancer outside of the intended treatment zone, defined as Gleason score 7 x < 10 years life expectancy
* Any medical condition that would compromise the subject's ability to safely ● Active bleeding disorder
* Use of coumadin or any other anticoagulant, unless anticoagulation can be temporarily reversed or stopped for a window of at least 7 days peri-procedure
* Active urinary tract infection x Active prostate abscess, prostatitis, or neurogenic bladder x Any prior treatment for prostate cancer, including:

  * Radical prostatectomy
  * Radiation therapy (external beam or brachytherapy)
  * Cryotherapy
  * High intensity focused ultrasound (HIFU) treatment o Photodynamic therapy o Androgen deprivation therapy
* Prior prostate, bladder neck, or urethral stricture surgery
* Any prostate debulking procedure, including: transurethral resection of prostate, photovaporization, or electrovaporization
* Transurethral incision of bladder neck x Urethral stricture dilation or reconstruction
* Use of 5-alpha reductase inhibitors within 6 months of treatment x Prior significant rectal surgery (hemorrhoidectomy is acceptable)
* Rectal fissure, fibrosis, stenosis, or other anatomic abnormality precluding insertion of transrectal device
* Inflammatory bowel disease x Urinary tract or rectal fistula x Previous urethral sling, artificial urinary sphincter or penile prosthesis surgery.
* Any contraindication to MRI (contrast allergy, severe claustrophobia, MRI-incompatible prosthesis, MRI-unsafe aneurysm clips)

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — eligibility based on physical existence of prostate.
Enrollment: 10 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety based on cumulative adverse events incurred | From treatment at 1 week, 1 month, and every 3 months until one year.
  Safety will be determined by the cumulative number, type, and severity of adverse events incurred by subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Pantuck, M.D., Principal Investigator — University of California at Los Angeles
Locations (1):
- University of California at Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No